CLINICAL TRIAL: NCT00881166
Title: Safety and Dose Finding Study of Oral MP470, a Multi-targeted Tyrosine Kinase Inhibitor, in Combination With Standard-of-Care Chemotherapy Regimens
Brief Title: Safety of MP470 in Combination With Standard-of-Care Chemotherapy Regimens to Treat Solid Tumors
Acronym: SGI-0470-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGI-0470-02
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Malignant Disease
Keywords: MP-470; Multi-targeted Tyrosine Kinase Inhibitor; Malignant disease
MeSH Terms: interventions — amuvatinib; Topotecan; Docetaxel; Erlotinib Hydrochloride; Paclitaxel; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): oral MP-470 + paclitaxel/carboplatin
  Interventions: Drug: MP-470 + paclitaxel/carboplatin
- 2 (Experimental): oral MP-470 + carboplatin/etoposide
  Interventions: Drug: MP-470 + carboplatin/etoposide
- 3 (Experimental): oral MP-470 + topotecan
  Interventions: Drug: MP-470 + topotecan
- 4 (Experimental): oral MP-470 + docetaxel
  Interventions: Drug: MP-470 + docetaxel
- 5 (Experimental): oral MP-470 + Erlotinib
  Interventions: Drug: MP-470 + erlotinib

INTERVENTIONS:
Drug: MP-470 + topotecan — Topotecan 1.5 mg/m2 IV infusion over 30 minutes on Days 1-5
  Arms: 3
Drug: MP-470 + docetaxel — Docetaxel 75 mg/m2 IV infusion over 1 hour on Day 1
  Arms: 4
Drug: MP-470 + erlotinib — 150 mg PO once daily at least 1 hour before or 2 hours after eating
  Arms: 5
Drug: MP-470 + paclitaxel/carboplatin — Paclitaxel 200 mg/m2 IV infusion over 3 hours followed by carboplatin IV infusion over 1 hour to a target AUC of 6 mg∙min/mL on Day 1
  Arms: 1
Drug: MP-470 + carboplatin/etoposide — Carboplatin IV infusion over 1 hour to target AUC of 5 mg min/mL on Day 1 followed by etoposide 100 mg/m2 IV infusion over 2 hours on Days 1-3
  Arms: 2

SUMMARY:
Adult subjects with malignant disease appropriate for treatment with carboplatin/paclitaxel, carboplatin/etoposide, topotecan, docetaxel or erlotinib according to the standard dosing regimen will be enrolled in each treatment arm.

Primary objective: Determine the MTD.

Secondary objectives: Response rates, PK, quantify MP-470 on PK of SOC, and collect pharmacodynamic information. Evaluate the overall safety of MP-470 when co-administered with specific SOC treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Malignant disease appropriate for initiating treatment with carboplatin/paclitaxel, carboplatin/etoposide, topotecan, docetaxel, or erlotinib.
2. Must be able to read, understand, and sign the IRB approved Informed Consent Form.
3. At least 18 years old.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Adequate bone marrow function; normal renal and hepatic function, normal cardiac function.

Exclusion Criteria:

1. Any other active invasive malignancy except non-melanoma skin cancers or cervical carcinoma in situ.
2. History of significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure and/or myocardial infarction.
3. Received any anticancer agent(s) within the past 3 weeks, including investigational agents, chemotherapy (6 weeks for nitrosoureas or mitomycin), immunotherapy, biologic or hormonal therapy other than LHRH agonists.
4. Received prior radiation therapy within the past 4 weeks.
5. Any serious, uncontrolled active infection that requires systemic treatment or known infection with HIV, HCV or HBV.
6. Patient requires treatment with immunosuppressive agents other than corticosteroids appropriate for the SOC chemotherapy regimen or those at stable doses for at least 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | March 2010

SECONDARY OUTCOMES:
Response rate | March 2010
Pharmacokinetics, pharmacodynamic effects on biomarker modulation. | March 2010
Experience DLT | March 2010

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Premiere Oncology, Scottsdale, Arizona
  - Premiere Oncology, Santa Monica, California
  - Audie Murphy Veterans Memorial Hospital (VA), San Antonio, Texas
  - CTRC at the UT Health Science Center at San Antonio, San Antonio, Texas
  - South Texas Accelerated Research Therapy (START), San Antonio, Texas

REFERENCES:
- [Derived] Mita M, Gordon M, Rosen L, Kapoor N, Choy G, Redkar S, Taverna P, Oganesian A, Sahai A, Azab M, Bristow R, Tolcher AW. Phase 1B study of amuvatinib in combination with five standard cancer therapies in adults with advanced solid tumors. Cancer Chemother Pharmacol. 2014 Jul;74(1):195-204. doi: 10.1007/s00280-014-2481-1. Epub 2014 May 22. PMID 24849582